CLINICAL TRIAL: NCT00191347
Title: A Phase II Study of Biweekly Pemetrexed and Gemcitabine in Patients With Metastatic Breast Cancer
Brief Title: A Study of Biweekly Pemetrexed and Gemcitabine in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9305; H3E-CA-S050
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: pemetrexed
Drug: gemcitabine

SUMMARY:
This study is designed to determine the efficacy of the biweekly pemetrexed/gemcitabine regimen when given to patients with metastatic breast cancer. Each agent has well demonstrated antitumor activity in patients with locally advanced or metastatic breast cancer. In addition, in the phase I combination trial of the two agents, a durable tumor response was seen in one out of three heavily pretreated breast cancer patients (Adjei et al. 2000). Therefore, it is reasonable to expect that the combination of pemetrexed and gemcitabine administered may be associated with considerably more anti-tumor activity than either agent alone. If such activity is seen in this study, randomized studies comparing this combination with other active agents or combinations of active agents will be considered.

ELIGIBILITY:
INCLUSION:

1. Have a performance status of 0 to 2 on the ECOG performance status schedule.
2. Patients may have had up to one prior systemic chemotherapy for metastatic disease is allowed. Prior adjuvant therapy is allowed if it has been more than one year since the end of therapy.
3. Patients must have measurable disease as defined by RECIST criteria (Therasse et al. 2000):
4. Have adequate organ function including the following

EXCLUSION:

1. Have serious concomitant systemic disorders (eg, active infection) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-10; Study Completion 2005-11

PRIMARY OUTCOMES:
To determine the objective tumor response rate for pemetrexed plus gemcitabine administered every 14 days, in patients with MBC who have received up to one prior chemotherapy for metastatic disease(not including prior adjuvant chemotherapy)

SECONDARY OUTCOMES:
To measure time-to-event efficacy variables including: time to objective tumor response for responding patients, duration of response for responding pts, time to treatment failure, time to progressive disease, progression free survival, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours,EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario, Canada